CLINICAL TRIAL: NCT05644236
Title: Safety and Efficacy Evaluation of Mouth Wash(Glister Mouth Wash): Pilot Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wonju Severance Christian Hospital (Other)
Responsible Party: Principal Investigator, Kyu Jae Lee, Professor, Wonju Severance Christian Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: EMB-2020-02; 2020-51-0447 (Other Grant/Funding Number: Amway Korea)
Record Dates: First submitted 2022-11-15; First posted 2022-12-09 (Actual); Last update posted 2022-12-09 (Actual); Status verified 2022-11

CONDITIONS: Oral Hygiene; Gingival Index; Cetylpyridinium Chloride
Keywords: mouthwash, cetylpyridinium chloride, oral hygiene
MeSH Terms: interventions — Mouthwashes

STUDY DESIGN:
Masking Description: Mouthwah solution was provided by sponsor who packed experimental and control solution in the bottle. Investigator and participants did not know the contents during treatment period.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- experimental group (Experimental): CPC-containing mouthwash solution
  Interventions: Other: mouthwash

INTERVENTIONS:
Other: mouthwash — After obtaining baseline information and randomizing the participants into two groups, dental scaling was performed, followed by clinical treatment. The participants were instructed to gargle twice daily for 7 days. All the participants were instructed not to eat or drink anything for at least 4 hours before the experiment. Oral hygiene, such as gargling and tooth brushing, was prohibited for 8 hrs before the visit.
  Other Names: Glister mouthwash

SUMMARY:
The goal of this clinical trial is to examine the efficacy of mouthwash containing 0.045% cetylpyridinium chloride (CPC) on oral health-related parameters] in [healthy conditions]. The main question[s] it aims to answer are:

* [ Trial 1: effect of immediate-use mouthwash containing CPC vs. non-CPC]
* [Trial 2: effect of concentrated-use mouthwash containing CPC vs. non-CPC] Participants will be treated by mouth wash 3 times a day for 4-weeks If there is a comparison group: Researchers will compare CPC containing mouthwash group and sham mouthwash groups treated with non CPC-containing mouthwash to see the effect of CPC on plaque index, mouth smell, gingival index and tongue coating index.

DETAILED DESCRIPTION:
2.1. Participants In all, 100 subjects were recruited to this clinical study according to the following inclusion criteria: i) Healthy male or female; ii) presence of >20 existing teeth (the number of remaining teeth); iii) no severe pathological soft tissue conditions, periodontitis, or extensive dental plaque; iv) Turesky modification of the Quigley-Hein Plaque Index (PI) of over 1.5 and Loe & Silness Gingival Index (GI) of over 1.5; vi) able to perform oral care/hygiene tasks on his/her own; vii) voluntary participation; and viii) willing to comply with the test protocol. Participants were excluded if they had any kind of visible or known disease requiring prophylactic antibiotic use.

2.2. Study design This was a randomized, controlled, double-blind clinical trial, and the intervention was gargling with the OR twice daily. The participants were randomly divided into four groups: control 1 (C1) (n=19), immediate-use CPC (IUC) (n=16), control 2 (C2) (n=19), and concentrated-use CPC (CUC) groups (n=19). Both C1 and C2 received ORs without CPC, whereas the experimental groups IUC and CUC received CPC ORs of different formulations (Amway Korea Ltd., Seoul, Republic of Korea). Randomized clinical trials (RCTs) are analyzed according to the intention-to-treat (ITT) principle and the per-protocol (PP) approach. ITT aims to assess the experimental design and PP analysis investigates the effect of receiving an assigned treatment. The participants underwent dental scaling before starting the intervention. Ethical approval was granted by the Institutional Research Ethics Review Board, Yonsei University, Wonju Severance Christian Hospital (IRBN CR321058) 2.3. Intervention After obtaining baseline information and randomizing the participants into two groups, dental scaling was performed, followed by clinical treatment. The participants were instructed to gargle twice daily for 7 days. All the participants were instructed not to eat or drink anything for at least 4 hours before the experiment. Oral hygiene, such as gargling and tooth brushing, was prohibited for 8 hours before the visit.

2.4. Measurment of H2S and methyl mercaptan, Quigley-Hein plaque index, Gingival Index,Tongue Coating Index.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male or female;
* presence of >20 existing teeth (the number of remaining teeth);
* no severe pathological soft tissue conditions, periodontitis, or extensive dental plaque;
* Turesky modification of the Quigley-Hein Plaque Index (PI) of over 1.5 and Loe & Silness Gingival Index (GI) of over 1.5; • able to perform oral care/hygiene tasks on his/her own;
* voluntary participation; and viii) willing to comply with the test protocol.

Exclusion Criteria:

* They excluded if they had any kind of visible or known disease requiring prophylactic antibiotic use.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2021-09-27 (Actual); Primary Completion 2021-11-30 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
hydrogen sulfide(H2S) and methyl mercaptan(CH3SH) | 4 weeks
  in the pretreatment versus post-treatment comparisons of the groups, levels of H2S (p < 0.01) and CH3SH (p < 0.01) were reduced significantly in cpc-containing mouthwash group (immediate-use and concentrated-use mouthwash) comparing non-CPC containing sham mouthwash.

SECONDARY OUTCOMES:
Quigley-Hein plaque index | 4 weeks
  the PI had decreased in all groups (Figure 3A). However, the IUC group showed significant antiplaque effects compared with the C1 group (p < 0.05). Improvement in periodontal health was seen 14 days after treatment, which was not observed in the CUC group (Figure 3B). Since OR without CPC also improved periodontal health, we further examined the group on day 28 of the trial. In addition, after 28 days, the CUC group showed antiplaque effects (p < 0.05). Overall, the IUC showed superior antiplaque activity and faster periodontal health-promoting effects than the CUC and control formulations.

OTHER OUTCOMES:
Gingival index | 4 weeks
  the highest increase in gingival health was observed 28 days after IUC administration (p < 0.05) (Figure 4A). Similar to the results for the PI, we did not observe significant changes in the gingival health of the C1 and C2 groups. As expected, gingival health improved significantly in the CUC group compared to in the C2 group, which was observed on study days 14 and 28 (Figure 4B).

CONTACTS AND LOCATIONS:
Overall Officials: Kyu-Jae Lee, Ph.D., Study Chair — Wonju College of Medicine, Yonsei University, Republic of Korea
Locations (1):
- Wonju Severance Christian Hospital, Wŏnju, Ganwon-do, South Korea

IPD SHARING:
Plan to Share IPD: No